CLINICAL TRIAL: NCT05851196
Title: Back to Back: the Forgotten Role of Back Muscle Characteristics to Tailor Exercise Therapy for Recurrent Non-specific Low Back Pain
Brief Title: The Forgotten Role of Back Muscle Characteristics to Tailor Exercise Therapy for Recurrent Non-specific Low Back Pain
Acronym: Back-to-Back
Status: Recruiting | Type: Observational
Sponsor: Hasselt University (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Principal Investigator, Lotte Janssens, Prof. Dr., Hasselt University
Other Study IDs: S67192
Record Dates: First submitted 2023-04-07; First posted 2023-05-09 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Low Back Pain; Back Pain Lower Back Chronic
Keywords: Proprioceptive postural control; Muscle volume; Muscle activation; Muscle oxygenation; Muscle fiber type composition; Proprioceptive training
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Muscle biopsies of the lumbar multifidus and erector spinae
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with non-specific low back pain: Individuals with chronic non-specific ow back pain
  Interventions: Other: Proprioceptive training
- Healthy controls: Healthy, age- and sex-matched individuals without low back pain

INTERVENTIONS:
Other: Proprioceptive training — A physiotherapist tailors the exercises to the patient's functional demands and pain- or fear-inducing activities. Guided by the therapist, patients look for ways to integrate the exercises into their daily life activities. Each week, patients receive feedback from the physiotherapist, and the training program is gradually progressed. The patients are instructed to perform the exercises daily, integrated into their daily activities, hobbies, and work. The program contains: (1) exercises to improve the sense of posture and movement, (2) exercises to correct the reference frame from which patients control posture and movement, (3) muscle control exercises, (4) exercises to increase variability in postures and movement patterns, (5) functionality: patients search for ways to correct and integrate alternative postures and movement patterns into their daily life, (6) high training frequency and high load, (7) focus on sensing, localizing and differentiating, rather than movement control.
  Groups: Patients with non-specific low back pain

SUMMARY:
Patients with non-specific low back pain will be compared to healthy, age- and sex-matched controls to determine the most discriminating back muscle characteristics and to delineate possible phenotypes of patients with non-specific low back pain showing impaired proprioceptive postural control. Additionally, the group of patients with non-specific low back pain will receive a 16-week, high-load proprioceptive training program. The effects of this training program on the different back muscle characteristics and proprioceptive postural control will be evaluated.

DETAILED DESCRIPTION:
The Back-to-Back study consists of a cross-sectional study and a proof-of-concept study. The cross-sectional study aims to gain more insight into the peripheral underlying mechanisms of impaired proprioceptive postural control in patients with non-specific low back pain. Macroscopic, microscopic, hemodynamic, and electrophysiological characteristics of the lumbar multifidus and erector spinae muscles will be compared between patients with non-specific low back pain and healthy, age- and sex-matched controls. The interrelatedness between these back muscle characteristics and the correlation with proprioceptive postural control will be examined. The most discriminating muscle characteristics will be determined based upon which phenotypes of patients with non-specific low back pain will be delineated. The proof-of-concept study aims to assess the effects of high-load proprioceptive training on back muscle characteristics and proprioceptive postural control in patients with non-specific low back pain.

ELIGIBILITY:
Inclusion Criteria:

Patients with non-specific low back pain:

* Aged 18-60 years
* Non-specific low back pain without radicular leg pain
* Mechanical low back pain with episodes of <4 on the numerical pain rating scale and episodes of >6 on the numerical pain rating scale
* Non-specific low back pain for three months or more
* Score of 20% or more on the Modified Low Back Pain Disability Questionnaire
* Informed consent to participate

Healthy controls:

* Aged 18-60 years
* No history of low back pain needing medical treatment or resulting in a limited activity level
* No low back pain in the previous six months
* Informed consent to participate

Exclusion Criteria:

* Pregnancy
* Previous trauma or surgery to the spine, pelvis or lower limbs
* Structural spinal deformity (e.g., scoliosis)
* Neurological, neuromuscular, respiratory or systemic disease
* Central sensitization: score of 50/100 or more on the Central Sensitization Inventory
* Specific vestibular or balance problems
* Acute lower limb or neck problems
* Body mass index of 30 kg/m² or more

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Flemish Brabant
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Proprioceptive postural control at baseline 1 (t= 0 weeks) | At baseline 1 (t= 0 weeks)
  Center-of-pressure displacement in response to ankle and/or back muscle vibration and the Relative Proprioceptive Weighting ratio will be calculated.
Proprioceptive postural control at baseline 2 (t= 8 weeks) (only for patients) | At baseline 2 (t= 8 weeks)
  Center-of-pressure displacement in response to ankle and/or back muscle vibration and the Relative Proprioceptive Weighting ratio will be calculated.
Proprioceptive postural control after 8 weeks of training (t= 16 weeks) (only for patients) | After 8 weeks of training (t= 16 weeks)
  Center-of-pressure displacement in response to ankle and/or back muscle vibration and the Relative Proprioceptive Weighting ratio will be calculated.
Proprioceptive postural control after 16 weeks of training (t= 24 weeks) (only for patients) | After 16 weeks of training (t= 24 weeks)
  Center-of-pressure displacement in response to ankle and/or back muscle vibration and the Relative Proprioceptive Weighting ratio will be calculated.
Proprioceptive postural control 16 weeks after the end of training (t= 40 weeks) (only for patients) | 16 weeks after the end of training (t= 40 weeks)
  Center-of-pressure displacement in response to ankle and/or back muscle vibration and the Relative Proprioceptive Weighting ratio will be calculated.
Macroscopic characteristiscs of the lumbar multifidus and erector spinae muscles at t= 0 weeks (only for healthy controls) | At t= 0 weeks
  Muscle volume and quality will be measured with 3D freehand ultrasound, muscle cross-sectional area and thickness will be evaluated with 2D ultrasound.
Macroscopic characteristiscs of the lumbar multifidus and erector spinae muscles at baseline 2 (t= 8 weeks) (only for patients) | At baseline 2 (t= 8w, 2nd baseline)
  Muscle volume and quality will be measured with 3D freehand ultrasound, muscle cross-sectional area and thickness will be evaluated with 2D ultrasound.
Macroscopic characteristics of the lumbar multifidus and erector spinae muscles after 16 weeks of training (t= 24 weeks) (only for patients) | After 16 weeks of training (t= 24 weeks)
  Muscle volume and quality will be measured with 3D freehand ultrasound, muscle cross-sectional area and thickness will be evaluated with 2D ultrasound.
Macroscopic characteristisc of the lumbar multifidus and erector spinae muscles 16 weeks after the end of training (t= 40 weeks) (only for patients) | 16 weeks after the end of training (t= 40 weeks)
  Muscle volume and quality will be measured with 3D freehand ultrasound, muscle cross-sectional area and thickness will be evaluated with 2D ultrasound.
Microscopic muscle characteristics of the lumbar multifidus and erector spinae muscles at t= 0 weeks (only for healthy controls) | At t= 0 weeks
  Fine-needle biopsies of the lumbar multifidus and erector spinae muscles will be acquired.
Microscopic muscle characteristics of the lumbar multifidus and erector spinae muscles at baseline 2 (t= 8 weeks) (only for patients) | At baseline 2 (t= 8 weeks)
  Fine-needle biopsies of the lumbar multifidus and erector spinae muscles will be acquired.
Microscopic muscle characteristics of the lumbar multifidus and erector spinae muscles after 16 weeks of training (t= 24 weeks) (only for patients) | After 16 weeks of training (t= 24 weeks)
  Fine-needle biopsies of the lumbar multifidus and erector spinae muscles will be acquired.
Microscopic muscle characteristics of the lumbar multifidus and erector spinae muscles 16 weeks after the end of training (t= 40 weeks) (only for patients) | 16 weeks after the end of training (t= 40 weeks)
  Fine-needle biopsies of the lumbar multifidus and erector spinae muscles will be acquired.
Hemodynamic muscle characteristics of the lumbar multifidus and erector spinae muscles at baseline 1 (t= 0 weeks) | At baseline 1 (t= 0 weeks)
  The Tissue Oxygenation Index will be recorded continuously with near-infrared spectroscopy during different functional postures (prone lying, usual sitting, usual standing, standing with the trunk bent 25° forward).
Hemodynamic muscle characteristics of the lumbar multifidus and erector spinae muscles at baseline 2 (t= 8 weeks) (only for patients) | At baseline 2 (t= 8 weeks)
  The Tissue Oxygenation Index will be recorded continuously with near-infrared spectroscopy during different functional postures (prone lying, usual sitting, usual standing, standing with the trunk bent 25° forward).
Hemodynamic muscle characteristics of the lumbar multifidus and erector spinae muscles after 8 weeks of training (t= 16 weeks) (only for patients) | After 8 weeks of training (t= 16 weeks)
  The Tissue Oxygenation Index will be recorded continuously with near-infrared spectroscopy during different functional postures (prone lying, usual sitting, usual standing, standing with the trunk bent 25° forward).
Hemodynamic muscle characteristics of the lumbar multifidus and erector spinae muscles after 16 weeks of training (t= 24 weeks) (only for patients) | After 16 weeks of training (t= 24 weeks)
  The Tissue Oxygenation Index will be recorded continuously with near-infrared spectroscopy during different functional postures (prone lying, usual sitting, usual standing, standing with the trunk bent 25° forward).
Hemodynamic muscle characteristics of the lumbar multifidus and erector spinae muscles 16 weeks after the end of training (t= 40 weeks) (only for patients) | 16 weeks after the end of training (t= 40 weeks)
  The Tissue Oxygenation Index will be recorded continuously with near-infrared spectroscopy during different functional postures (prone lying, usual sitting, usual standing, standing with the trunk bent 25° forward).
Electrophysiological muscle characteristics of the lumbar multifidus and erector spinae at baseline 1 (t= 0 weeks) | At baseline 1 (t= 0 weeks)
  Muscle activitation levels and patterns will be measured with surface electromyography during different functional postures (prone lying, usual sitting, usual standing, standing with the trunk bent 25° forward).
Electrophysiological muscle characteristics of the lumbar multifidus and erector spinae at baseline 2 (t= 8 weeks) (only for patients) | At baseline 2 (t= 8 weeks)
  Muscle activitation levels and patterns will be measured with surface electromyography during different functional postures (prone lying, usual sitting, usual standing, standing with the trunk bent 25° forward).
Electrophysiological muscle characteristics of the lumbar multifidus and erector spinae after 8 weeks of training (t= 16 weeks) (only for patients) | After 8 weeks of training (t= 16 weeks)
  Muscle activitation levels and patterns will be measured with surface electromyography during different functional postures (prone lying, usual sitting, usual standing, standing with the trunk bent 25° forward).
Electrophysiological muscle characteristics of the lumbar multifidus and erector spinae after 16 weeks of training (t= 24 weeks) (only for patients) | After 16 weeks of training (t= 24 weeks)
  Muscle activitation levels and patterns will be measured with surface electromyography during different functional postures (prone lying, usual sitting, usual standing, standing with the trunk bent 25° forward).
Electrophysiological muscle characteristics of the lumbar multifidus and erector spinae 16 weeks after the end of training (t= 40 weeks) (only for patients) | 16 weeks after the end of training (t= 40 weeks)
  Muscle activitation levels and patterns will be measured with surface electromyography during different functional postures (prone lying, usual sitting, usual standing, standing with the trunk bent 25° forward).

SECONDARY OUTCOMES:
Disability due to low back pain | Controls: once, immediately after inclusion, Patients: 5 times, immediately after inclusion (t= 0w), after 8 weeks (t= 8w, 2nd baseline), after 8 weeks of training (t= 16w), after 16 weeks of training (t= 24w), 16 weeks after the end of training (t= 40w)
  Participants will be asked to complete the Modified Low Back Pain Disability Questionnaire.
Risk for future work disability due to low back pain | Controls: once, immediately after inclusion, Patients: 5 times, immediately after inclusion (t= 0w), after 8 weeks (t= 8w, 2nd baseline), after 8 weeks of training (t= 16w), after 16 weeks of training (t= 24w), 16 weeks after the end of training (t= 40w)
  Participants will be asked to complete the short version of the Örebro Musculoskeletal Pain Screening Questionnaire
Pain-related fear of movement | Controls: once, immediately after inclusion, Patients: 5 times, immediately after inclusion (t= 0w), after 8 weeks (t= 8w, 2nd baseline), after 8 weeks of training (t= 16w), after 16 weeks of training (t= 24w), 16 weeks after the end of training (t= 40w)
  Participants will be asked to complete the Tampa Scale for Kinesiophobia.
Fear-avoidance beliefs about physical activity and work | Controls: once, immediately after inclusion, Patients: 5 times, immediately after inclusion (t= 0w), after 8 weeks (t= 8w, 2nd baseline), after 8 weeks of training (t= 16w), after 16 weeks of training (t= 24w), 16 weeks after the end of training (t= 40w)
  Participants will be asked to complete the Fear-Avoidance Beliefs Questionnaire.
Pain catastrophizing | Controls: once, immediately after inclusion, Patients: 5 times, immediately after inclusion (t= 0w), after 8 weeks (t= 8w, 2nd baseline), after 8 weeks of training (t= 16w), after 16 weeks of training (t= 24w), 16 weeks after the end of training (t= 40w)
  Participants will be asked to complete the Pain Catastrophizing Scale.
Anxiety and depression | Controls: once, immediately after inclusion, Patients: 5 times, immediately after inclusion (t= 0w), after 8 weeks (t= 8w, 2nd baseline), after 8 weeks of training (t= 16w), after 16 weeks of training (t= 24w), 16 weeks after the end of training (t= 40w)
  Participants will be asked to complete the Hospital Anxiety and Depression Scale.
Habitual physical activity | Controls: once, immediately after inclusion, Patients: 5 times, immediately after inclusion (t= 0w), after 8 weeks (t= 8w, 2nd baseline), after 8 weeks of training (t= 16w), after 16 weeks of training (t= 24w), 16 weeks after the end of training (t= 40w)
  Participants will be asked to complete the Baecke Questionnaire.

OTHER OUTCOMES:
Age | Immediately after inclusion
  Age (years) will be recorded.
Sex (male/female) | Immediately after inclusion
  Sex will be recorded.
Highest level of education | Immediately after inclusion
  Highest level of education will be recorded.
Current employment status | Immediately after inclusion
  Current employment status will be recorded.
Body weight (kg) | Immediately after inclusion
  Body weight (kg) will be recorded.
Height (cm) | Immediately after inclusion
  Height (cm) will be recorded.
Handedness (left, right) | Immediately after inclusion
  Handedness will be recorded.
Current pain intensity (only for patients) | Immediately after inclusion
  Patients will be asked to rate the current intensity of pain in their lower back (and leg if present) on a Numerical Rating Scale with anchors 0= no pain and 10= worst pain.
Duration of low back pain (only for patients) | Immediately after inclusion
  The duration of low back pain (months) will be recorded.
Medication use (only for patients) | Immediately after inclusion
  Medication use will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Lotte Janssens, PhD, Principal Investigator — Hasselt University
Locations (2):
- Belgium (2):
  - REVAL Rehabilitation Research Center, Hasselt University, Diepenbeek
  - Department of Rehabilitation Sciences, KU Leuven, Leuven

IPD SHARING:
Plan to Share IPD: No